CLINICAL TRIAL: NCT04650685
Title: Anti-Plaque and Anti-Gingivitis Effectiveness of the Newly Invented Salvadora Persica Toothbrush Compared to Salvadora Persica Chewing Stick: A Randomised Controlled Trial
Brief Title: Effectiveness of Salvadora Persica Miswak in Improving Plaque Control and Gingival Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, :Nurulhuda Mohd, Principal investigator; Lecturer and Clinical Consultant (Periodontist), National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UKM PPI/111/8/JEP-2020-620
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Gingivitis; Dental Plaque
Keywords: Miswak; Dental biofilms; Periodontal disease
MeSH Terms: conditions — Gingivitis; Dental Plaque; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Group 1: Salvadora persica toothbrush (under the brand of Al-Abyad) that is to be used without toothpaste application.
  Group 2: Salvadora persica chewing sticks (under the brand of Al-Khair) with uniform diameter (1cm) and equal length of 15 cm. Three miswak chewing sticks will be distributed to each participant (one stick/week). Upon receiving, they will be sealed in air-tight plastic bags. This miswak chewing stick is also to be used without the application of any toothpaste.
  Group 3: Participants will be given a regular, standard straight-handle soft-bristle Colgate toothbrush each to be used with the application of Colgate® fluoride toothpaste.
  Professional cleaning of scaling and polishing will be performed if needed during the first visit.
Who Masked: Outcomes Assessor
Masking Description: A research assistant will be responsible for randomisation and grouping hence the outcome assessor will not be aware of which group the participant belonged to. One outcome assessor will be responsible for the clinical evaluations, who will be masked to the intervention groups throughout the study. Individual participants will not be informed about the study hypothesis and will strictly be asked not to disclose to the outcome assessor which oral hygiene tool they are using. This is to ensure the outcome assossor is fully blinded in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The novel Salvadora persica toothbrush (Experimental): The novel toothbrush is under Al-Abyad Miswak brand that will be supplied by Insight Prestige Sdn Bhd. Participants are expected to use this oral hygiene tool for 3 weeks.
  Interventions: Device: The novel Salvadora persica toothbrush
- The Salvadora persica (miswak) chewing sticks (Experimental): The chewing sticks are under the brand of Al-Khair. They will be prepared into equal length of 15 cm with uniform diameter of 1.0-1.5 cm and are sealed in airtight plastic bags. Participants are expected to use this oral hygiene tool for 3 weeks.
  Interventions: Device: The Salvadora persica (miswak) chewing stick
- Standard toothbrush and toothpaste (control) (Other): Participants will be given straight-handle soft-bristle Oral-B™ standard toothbrush and Colgate® fluoride tooth. Participants are expected to use this oral hygiene tool for 3 weeks.
  Interventions: Device: Standard toothbrush and toothpaste (control)

INTERVENTIONS:
Device: The novel Salvadora persica toothbrush — The novel Salvadora persica toothbrush will be used twice daily without the application of toothpaste. Modified bass technique will be applied. A demonstration by another investigator will be done via video, written instructions and a tell-show-do method using typodont model.
  Arms: The novel Salvadora persica toothbrush
Device: The Salvadora persica (miswak) chewing stick — The Salvadora persica chewing stick will be used twice daily without the application of toothpaste. The Salvadora persica chewing sticks need to be prepared prior to use. A five-finger grip technique will be applied. A demonstration by another investigator will be done via video, written instructions and a tell-show-do method using typodont model.
  Arms: The Salvadora persica (miswak) chewing sticks
Device: Standard toothbrush and toothpaste (control) — The novel Salvadora persica toothbrush will be used twice daily without the application of toothpaste. Modified bass technique will be applied. A demonstration by another investigator will be done via video, written instructions and a tell-show-do method using typodont model.
  Arms: Standard toothbrush and toothpaste (control)

SUMMARY:
Dental plaque is a main etiologic agent in periodontal disease. Global of Burden Disease Study 2016 ranked periodontal disease as the 11th most prevalent disease affecting 10.5% population worldwide. Tooth brushing is a reliable mechanical means to control dental plaque accumulation in order to maintain oral health. For decades, studies have demonstrated the efficiency of unprocessed Salvadora persica (miswak) chewing stick practice as an alternative to a standard toothbrush. Recently, a local Malaysian company has invented and successfully mass manufactured a world-first Salvadora persica toothbrush where its nylon bristles are primarily mixed with miswak powder and natural silica. With the benefits of Salvadora persica properties intact, it is also claimed to be effective without the application of toothpaste. However, the claim remains to be fully elucidated. There is also no randomized controlled trial available evaluating the efficacy of Salvadora persica toothbrush to date. Therefore, the aim of this study is to evaluate the effectiveness of the newly invented Salvadora persica toothbrush on oral health, particularly on anti-plaque and anti-gingivitis effects. The patient related-outcomes of Salvadora persica on a short-term use will also be assessed. The hypotheses of this study are that Salvadora persica toothbrush does not contribute to the significant effects on oral health and there is no difference in the use of Salvadora persica chewing stick, Salvadora persica toothbrush as well as the standard toothbrush on anti-plaque and anti-gingivitis in a standardized manner. Additionally, a hypothesis that there is no patient-related outcome of Salvadora persica on a short-term use has also been devised. A randomized, single blind, and parallel clinical study will be conducted over a five-week period involving the healthy non-dental students of the National University of Malaysia. This study consists of three groups of different oral hygiene tools: (i) Salvadora persica toothbrush; (ii) Salvadora persica chewing stick; and (iii) Standard toothbrush and toothpaste as control. The primary outcomes of this study are the clinical parameters that will be recorded at four different appointments. Salvadora persica toothbrush is expected to show positive effects to that of standard toothbrush with respect to plaque and gingivitis control. This study is thus designed to provide an insight on Salvadora persica toothbrush as a good preventive home care therapy.

DETAILED DESCRIPTION:
The specific objectives of this clinical trial are to evaluate and compare the oral health status on gingivitis and plaque control in a standardised manner between Salvadora persica toothbrush and Salvadora persica chewing stick usage, to investigate the clinical efficiency of Salvadora persica toothbrush and Salvadora persica chewing stick on plaque removal in comparison with standard toothbrush, and to assess the patient-related outcome of Salvadora persica on a short-term use. A 20% drop out rate is to be expected.

Convenience sampling will be used in this study involving non-dental students of the National University of Malaysia Kuala Lumpur Campus. They are within the radius of the study site therefore are easy to obtain. Their manual dexterity and attitude towards oral health are the critical basis needed to maintain proper oral cleanliness, hence justified this non-probability sampling method selected.

The sample size calculation formula will be devised from a pilot study, which will primarily be conducted first involving five participants on each arm who are selected by a convenience sampling. The mean and standard deviation of two clinical parameters; Gingival Index and Plaque Index of the three groups assigned will be calculated. A confidence level of 95% with margin of error of 0.5 will be set to calculate the appropriate sample size for this study. The calculated sample size will be raised to the nearest 5 e.g. 23 will be increased to 25, to improve the validity of the study.

Prior to the participants' recruitment, the information sheet and the consent forms will be distributed. Enough time will be given for them to read and understand the study protocol before they agree to participate in this study. Those who give a consent to involve in the study will be enrolled as the participants. The principal investigator must ensure the participants understand the benefits and risks of the study. This information will be conveyed in an objective manner and any queries from the participants will be answered truthfully. The participants will have the right to refuse in participating in this study.

In this study, one principal examiner will be involved for the clinical evaluations. Prior to the initiation of the study, the examiner will be calibrated to measure the clinical parameters of periodontal attachment level, Plaque Index, and Gingival Index against another researcher who will act as a benchmark. For the assessment of intra-examiner reliability, these three clinical parameters will be recorded on five non-dental students who are not participating in this study, under the same circumstances with similar patient positioning, light positioning, and instruments. A weighted kappa score will be used to calculate the strength of agreement for both inter-examiner and intra-examiner reliability. An agreement is achieved when the values are >0.8.

The clinical protocol will be conducted over a five-week period, with a total of 4 clinical appointments performed throughout the study. In appointment 1 (baseline period), all subjects will be undergoing a clinical examination prior to participating in the study. Subjects will also be interviewed using a structured questionnaire to assess their oral hygiene habits i.e. frequency and methods of toothbrushing, frequency of dental visits, as well as history of adjunct oral hygiene aid e.g. floss, and mouthwash. To ensure that all included subjects received the same standard of care, all participants will receive professional dental cleaning consisting of scaling and polishing during the first visit.

During appointment 2 (pre-intervention period), the proper technique of using the designated standard and the new miswak toothbrushes, as well as miswak chewing sticks will be explained both verbally and visually using models to each participant accordingly by another trained dentist who is blinded to the study protocol. In addition, all subjects received written instructions with coloured pictures demonstrating the modified bass technique for tooth brushing. Subjects who are selected to use miswak chewing stick will be given a sheet of written instructions demonstrating the proper preparation and preservation techniques of miswak chewing stick. It is very crucial that the participants are reminded to avoid using other means of cleaning devices, dentifrices, or adjuncts for the following three weeks of the study. Participants are also encouraged to seek for oral hygiene reinforcement wherever they feel the need to do so throughout the study period. At this visit, participants will also be asked to answer the pre-intervention S-OHIP questionnaires in front of an interviewer, which has also been validated both in English and Malay versions.

Appointment 3 is one-week post-intervention while appointment 4 will be three weeks post-intervention. In these visits, clinical examination will be carried out and assessment of any adverse effects of oral hygiene tools used will be taken. At final visit (appointment 4), participants will be asked to answer the post-intervention S-OHIP questionnaires in front of an interviewer.

Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 26 (SPSS Inc., Chicago, IL, USA). For the primary outcomes measure, the values for Plaque Index and Gingival Index will be expressed as mean ± standard deviation. These parametric variables will be analysed using Kruskal-Wallis test to determine whether significant differences exist between the three independent groups from baseline to pre-intervention, and from pre-intervention to first and third week of analysis of post-intervention. Statistical significance will be set at the 95% confidence level (α=0.05) for hypothesis testing. Post-hoc tests for multiple comparison of significant mean differences between groups at specific time intervals will be performed with either Dunn-Bonferroni Test (less statistical powerful and conservative) or several Mann-Whitney U Test (inflation of Type I error), with the understanding of both test limitations. For the secondary outcome measures, frequencies and percentages will be used to describe the distribution of responses for each question in OHIP-14 questionnaires. Depending on the distribution the data later, independent sample t-test/ANOVA or the Mann-Whitney/Kruskal-Wallis tests will be used to assess the median OHIP-14 scores based on sample characteristics, oral hygiene habits/practices and oral status. Meanwhile, the comparisons of all groups for the presence and frequency of both objective and subjective adverse reactions (nominal values) will be tested with Chi-Square or Fisher's exact test where appropriate. Analysis of the subjective and objectives adverse events sessions will be done using McNemar test.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are systemically healthy
2. Individuals who have ≥ 24 teeth
3. Individuals who have Basic Periodontal Examination score 0, 1 and 2 only with no periodontal deep pocket more than 5.5mm (gum disease)
4. Individuals who have never smoke cigarettes or other tobacco products

Exclusion Criteria:

1. Individuals who are the habitual users of miswak chewing sticks, or have experienced in using them
2. Individuals who wear orthodontic appliances (braces)
3. Individuals who have grossly decayed teeth, gross overhanging restorations, severe malpositioned teeth (crowded teeth) and/or gingival recession (receding gum), have crowns placed, and wear partial dentures
4. Individuals who have current or previous history of periodontal treatment (gum treatment) including root surface debridement/periodontal surgery
5. Individuals who are poor in manual dexterity
6. Individuals who are pregnant or lactating mothers
7. Individuals who have taken antibiotics in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Probing attachment level | 5 weeks
  Firstly, the periodontal pocket depth (PPD) will be assessed at six points per tooth. The measurement will be performed using a University of North Carolina probe (PCP-UNC 15) probe, which has a clear black coding of every millimetre demarcation that is up to 15 mm length.
  Then, probing attachment level will be assessed to the nearest millimetre by the same probe and expressed as the distance in millimetres from the cemento-enamel junction (CEJ) to the base of the pocket. This clinical assessment requires the measurement of the distance from the CEJ to the free gingival margin (FGM) for all six points. Periodontal attachment level is calculated by subtracting the distance of the CEJ to the FGM from the PPD. However, because gingival recession is an exclusion criterion in this study, gingival margin might be located at the CEJ at baseline, hence periodontal attachment level might be of similar value with to PPD.
Gingival Index | 5 weeks
  This implies the gingival status by the examination of the severity of gingival inflammation. In addition, the initiation of bleeding will be noted by gently stroking the entrance to the gingival sulcus with a blunt periodontal probe.
  Scores of 0, 1, 2 and 3 will be given. The explanation of the scores are as follows:
  0 = Absence of plaque
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface, not visible by the naked eye
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface
Plaque Index | 5 weeks
  Before the presence of dental plaque level is examined, the disclosing solution will be applied on the small cotton swab and then gently dabbed on the tooth surface. The participants will be instructed not to rinse their mouth with water until the examination is completed.
  Scores of 0, 1, 2 and 3 will be given. The explanation of the scores are as follows:
  0 = Absence of plaque
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface, not visible by the naked eye
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be by the naked eye
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface

SECONDARY OUTCOMES:
S-OHIP(M) scores | 3 weeks
  This oral health-related quality of lifeparameter will be measured using the translated and validated short version questionnaires of the Malaysian Oral Health Impact Profile, designated as S-OHIP(M). These questionnaires are patient-centred outcome measures that assess the patient's responses to the various oral health indicators. It has 14 items grouped into seven domains: namely functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses are coded using a 5-point Likert scale: 0 = never; 1 = seldom; 2 = sometimes; 3 = quite often; and 4 = very often. A high score indicates poor OHR-QoL, while the total number of patients choosing "never" and "seldom" represents the percentage of patients with satisfactory OHR-QoL.
  Participants are expected to be able to read and understand Malay and/or English.
Prevalence of subjective and objective evaluation of adverse events on oral hygiene tool use | 3 weeks
  These adverse events will be divided into two, namely the subjective assessment (self-reported adverse outcomes, if any, and the objective assessment (clinical assessment), which be performed to check for tissue irritations and discoloration and will be recorded as present/absent.

CONTACTS AND LOCATIONS:
Overall Officials: Nurulhuda Mohd, DDS, Principal Investigator — Department of Restorative Dentistry, Faculty of Dentistry, National University of Malaysia
Locations (1):
- Department of Restorative Dentistry, Faculty of Dentistry, National University of Malaysia, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Pihlstrom BL. Measurement of attachment level in clinical trials: probing methods. J Periodontol. 1992 Dec;63(12 Suppl):1072-7. doi: 10.1902/jop.1992.63.12s.1072. PMID 1479528
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Saub R, Locker D, Allison P. Derivation and validation of the short version of the Malaysian Oral Health Impact Profile. Community Dent Oral Epidemiol. 2005 Oct;33(5):378-83. doi: 10.1111/j.1600-0528.2005.00242.x. PMID 16128798
- [Background] Gibson JA, Wade AB. Plaque removal by the Bass and Roll brushing techniques. J Periodontol. 1977 Aug;48(8):456-9. doi: 10.1902/jop.1977.48.8.456. PMID 269253
- [Background] Poyato-Ferrera M, Segura-Egea JJ, Bullon-Fernandez P. Comparison of modified Bass technique with normal toothbrushing practices for efficacy in supragingival plaque removal. Int J Dent Hyg. 2003 May;1(2):110-4. doi: 10.1034/j.1601-5037.2003.00018.x. PMID 16451532
- [Background] Al-Otaibi M, Al-Harthy M, Gustafsson A, Johansson A, Claesson R, Angmar-Mansson B. Subgingival plaque microbiota in Saudi Arabians after use of miswak chewing stick and toothbrush. J Clin Periodontol. 2004 Dec;31(12):1048-53. doi: 10.1111/j.1600-051X.2004.00618.x. PMID 15560804
- [Background] Almas K, al-Lafi TR. The natural toothbrush. World Health Forum. 1995;16(2):206-10. No abstract available. PMID 7794468
- [Derived] Azizan NF, Mohd N, Nik Azis NM, Baharin B. Effectiveness of Salvadora persica toothbrush and Salvadora persica chewing stick in plaque and gingivitis control: a randomized control trial. BMC Complement Med Ther. 2023 Dec 14;23(1):456. doi: 10.1186/s12906-023-04295-z. PMID 38098022
- See also: The Good Practitioner's Guide to Periodontology — https://www.bsperio.org.uk/assets/downloads/good_practitioners_guide_2016.pdf